CLINICAL TRIAL: NCT00986336
Title: A Comparative Study of the Steady-state Pharmacokinetics of Risperidone and Topiramate on Monotherapy and During Combination Therapy in Patients With Bipolar or Schizoaffective Disorder
Brief Title: A Pharmacokinetic Study of Risperidone and Topiramate Administered Alone and in Combination in Patients With Bipolar Disorder or Schizoaffective Disorders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Senior Director, Clinical Leader - topiramate, Johnson & Johnson Pharmaceutical Research and Development, L.L.C.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR002857
Record Dates: First submitted 2009-09-25; First posted 2009-09-29 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-04

CONDITIONS: Bipolar Disorder
Keywords: topiramate; risperidone, bipolar disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Topiramate; Risperidone

ARMS (4):
- 001 (Experimental)
  Interventions: Drug: topiramate
- 002 (Experimental)
  Interventions: Drug: topiramate
- 003 (Experimental)
  Interventions: Drug: topiramate
- 004 (Experimental)
  Interventions: Drug: risperidone

INTERVENTIONS:
Drug: topiramate — 1-25 mg plus 1-100 mg tablet twice daily for 2 weeks (250 mg/day)
  Arms: 002
Drug: topiramate — 2-100 mg tablets twice daily for 2 weeks (400 mg/day)
  Arms: 003
Drug: risperidone — Twice daily, individualized dosing to stabilization at 1-6 mg/day.
  Arms: 004
Drug: topiramate — 2-25 mg tablets twice daily for 2 weeks (100 mg/day)
  Arms: 001

SUMMARY:
The purpose of this study is to assess the potential pharmacokinetic (absorption, distribution and excretion of the drug by the body) interaction between, and the safety of, topiramate and risperidone administered in combination in patients with a history of either bipolar spectrum or schizoaffective (bipolar type) disorders as defined by DSM-IV criteria.

DETAILED DESCRIPTION:
This was an open-label (both the investigator and the patient knew the identity of the study drug), nonrandomized pharmacokinetic (PK) study evaluating the interaction of topiramate and risperidone in patients with bipolar disorder. The study enrolled a sufficient number of patients to obtain 24 completed patients. Patients were men or women aged 18 to 55 years, inclusive, with a diagnosis of Bipolar Spectrum or Schizoaffective Disorder, who were not in the midst of an acute episode, and had not experienced an acute manic, major depressive, or schizoaffective episode for a minimum of 30 days prior to screening (enrollment was monitored to ensure that at least one-third of the study sample was of the same sex.) The study consisted of a screening phase and 3 treatment periods. In Period I, patients were stabilized to a clinically appropriate dose of risperidone within the range of 1 to 6 mg/day, administered in divided doses every 12 hours during a 2- to 3-week period (or longer as clinically necessary). Upon risperidone stabilization, serial blood and urine samples were obtained through 12 hours postdose for estimation of risperidone and its metabolite 9-OH-risperidone (metabolites are formed by metabolism of the drug) concentrations in Period I. In Period II, which lasted up to 6 weeks or longer as clinically necessary, topiramate was gradually escalated to 3 steady-state target doses, while risperidone therapy continued unchanged. There were up to 3 PK sampling periods (days when multiple blood and urine samples are taken to estimate the amount of topiramate and /or risperidone and its metabolite 9-OH-risperidone in blood or urine) when the patient achieved steady state at 100 mg/day topiramate (consistent amount of drug in blood with each dose); when/if the patient achieved steady state at 250 mg/day topiramate or maximum tolerated dose (MTD); and when/if the patient achieved steady state at 400 mg/day topiramate or MTD. During each PK sampling visit in Period II, serial blood and urine samples were obtained through 12 hours postdose for estimation of risperidone, 9-OH risperidone, and topiramate concentrations. In Period III, risperidone was gradually tapered while the 400-mg/day dose (or MTD) of topiramate was maintained. There were 2 PK sampling visits: when patients had attained steady state at a dose of 50% of the maximal risperidone dose reached in Period I; and when risperidone was discontinued for 7 days and patients were maintained on topiramate 400 mg/day or their respective MTD. During each PK sampling visit in Period III, serial blood and urine samples were obtained through 12 hours postdose for estimation of risperidone, 9-OH risperidone, and topiramate concentrations. Period I (risperidone stabilization): risperidone 1-6 mg/day for 2 to 3 weeks. Period II (topiramate dose escalation): topiramate administered for approximately 6 weeks titrated up to 3 potential target doses (100 mg/day, 250 mg/day and 400 mg/day), and risperidone continues unchanged. Period III (risperidone dose reduction): risperidone dose tapered to zero over a 4-week period while topiramate maintained at the target dose of 400 mg/day (or MTD).

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting DSM-IV criteria for either Bipolar I Disorder, Bipolar II Disorder, Cyclothymic Disorder, Bipolar Disorder NOS, or Schizoaffective Disorder (bipolar type)
* Patients not in the midst of an acute manic, major depressive, or schizoaffective episode and had not experienced an acute episode within the month prior to screening
* Women were to be postmenopausal for at least 1 year, or surgically incapable of childbearing, or practicing an acceptable method of birth control (hormonal contraception, intrauterine device, or barrier with spermicide were acceptable) and not pregnant at baseline.

Exclusion Criteria:

* Patients with a history of an acquired or hereditary neurologic disease, e.g., epilepsy or significant brain trauma
* Patients using prescription medication, including psychotropic medications, within 14 days prior to the first day of Period I with the exception of hormonal contraceptives (women), risperidone, or other medications approved by the sponsor
* Patients on depot medications (including but not limited to haloperidol decanoate)
* Patients who had taken acetazolamide, zonisamide, triamterene, dichlorphenamide, chronic antacids, or calcium supplements, or any medication associated with nephrolithiasis in the month prior to beginning TPM titration.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2001-02; Study Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the potential pharmacokinetic interaction between topiramate and risperidone in patients with bipolar disorder or schizoaffective disorders. | At each sampling visit during Periods I, II and III, blood and urine collected pre-morning dose and over a period of 12 hours post-dose.

SECONDARY OUTCOMES:
Assess the safety of multiple doses of topiramate in combination with varying doses of risperidone | At each sampling visit during Periods I, II and III

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A comparative study of the steady-state pharmacokinetics of risperidone and topiramate on monotherapy and during combination therapy in subjects with bipolar or schizoaffective disorders — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=493&filename=CR002857_CSR.pdf